CLINICAL TRIAL: NCT05528744
Title: Delineating the Molecular Spectrum and the Clinical, Imaging and Neuronal Phenotype of Chopra-Amiel-Gordon Syndrome
Status: Recruiting | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Maya Chopra, Director of Translational Genomic Medicine, Rosamund Stone Zander Translational Neuroscience Centre at Boston Children's Hospital, Boston Children's Hospital
Other Study IDs: P00041124
Record Dates: First submitted 2022-05-03; First posted 2022-09-06 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Genetic Disease; Chopra-Amiel-Gordon Syndrome; CAGS; ANKRD17
Keywords: Syndrome; Neurodevelopmental; ANKRD17 Loss of function; ANKRD17; Rare Disease
MeSH Terms: conditions — Genetic Diseases, Inborn; Syndrome; Rare Diseases | interventions — Observation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Biospecimen Retention: Samples With DNA — Human blood and skin samples for repository and the establishment of iPSC lines.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Proband: Study participants who have suspected or confirmed CAGS based on having a variant of uncertain significance, likely pathogenic variant, or pathogenic variant in ANKRD17 and clinical features of the condition.
  Interventions: Other: Observational Study
- Unaffected family members: Family members of the proband who do not have an ANKRD17 variant.
  Interventions: Other: Sample collection only

INTERVENTIONS:
Other: Observational Study — No intervention. This is an observational study
  Groups: Proband
Other: Sample collection only — Collection of blood and/or skin samples.
  Groups: Unaffected family members

SUMMARY:
The purpose of this study is to establish a registry of individuals with confirmed or suspected Chopra-Amiel-Gordon Syndrome (CAGS) to learn more about the range of symptoms, changes in the structure of the brain seen on imaging, and learning difficulties that individuals with this disorder may experience. The investigators will obtain medical history, family history, MRI records, patient photographs, and genetic test results from individuals with confirmed or suspected CAGS. A subset of participants will also undergo a standardized neurobehavioral assessment. This data will be maintained on a secure research database. Sample collection will be offered to participants for the functional testing and the generation of iPSC cell lines, for neuronal reprogramming and phenotyping.

DETAILED DESCRIPTION:
Heterozygous loss of function variants in ANKRD17 were recently implicated in a newly-identified rare intellectual disability syndrome. In an international collaborative effort spanning 4 years, the mutational and phenotypic spectrum of 34 patients were described (Chopra et al AJHG 2021). The core phenotypic features of this syndrome were shown to be intellectual disability, particularly affecting speech, and shared dysmorphic features. Variably present neurodevelopmental features were epilepsy /abnormal EEG, autism spectrum disorder, gait / balance difficulties and neuroimaging abnormalities. Extra-neurological features include growth delay, renal anomalies, hypermobility, pigmentary lesions and feeding problems. All variants were identified on whole exome or whole genome sequencing, and most were shown to be de novo and truncating, although some patients harbored missense variants particularly in highly conserved ankyrin repeat domains. While this initial project presented compelling evidence for a novel gene-disease relationship and established the key phenotypic features of this new disorder, there were limitations to this work. The neurodevelopmental profile and MRI findings were ascertained through physician report only rather than independent standardized assessment. Intriguingly, while it was observed that expressive language delay was more markedly affected than other developmental parameters, this observation was not validated with standardized patient evaluation. Currently, the impact of ANKRD17 haploinsufficiency on human neuronal morphology / excitability, and in turn, the correlation of this neuronal phenotype to the clinical neurodevelopmental profile is unknown. With this study, the investigators plan to deeply characterize the spectrum of clinical, neuroimaging and neuronal cellular features of this disorder, pairing preclinical with clinical science. The robust systematic evaluation of patients who are known or suspected to have this condition will lead to a better understanding of the true phenotypic spectrum and correlations to genotype. The inclusion of patients suspected to have CAGS, in particular, may expand the phenotypic and genotypic spectrum of the condition, and clarify diagnoses for these participants. This cross-sectional data will lay the foundations for the design of longitudinal studies and development of clinical trial endpoints. The generation of patient-specific iPSC lines and isogenic controls will allow for future projects to generate neuronal populations from clinically characterized patients, which will bridge the knowledge gap on the biological underpinnings of the disorder and potentially lead to biomarkers that reflect specific disrupted neurodevelopmental pathways.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a known or suspected diagnosis of CAGS
* Participants with a known diagnosis or CAGS have a disease-causing (likely pathogenic or pathogenic) variant in ANKRD17 evidenced by a pre-existing clinical genetic report.
* Participants with a suspected diagnosis of CAGS must have a variant of uncertain significance in CAGS evidenced by a pre-existing clinical genetic report and clinical features of CAGS

Exclusion Criteria:

* No evidence of a disease-causing or potentially disease-causing variant ANRKD17 variant on a pre-existing clinical genetic report.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population consists of patients of all ages and genders with a confirmed or suspected diagnosis of CAGS confirmed by pre-existing clinical genetic testing
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-08-27 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Research registry of molecular and phenotypic information related to CAGS | 4-5 years
  The primary endpoint of this cross-sectional natural history study will be the creation and implementation of a research registry of molecular and phenotypic information for CAGS.
Generation of patient-derived iPSC cell lines | 4-5 years
  An additional objective of this cross-sectional natural history study will be the generation of patient-derived iPSC cell lines. iPSC cell lines will be created from blood and skin samples of individuals with ANKRD17 variants, using samples from unaffected family members as controls.

CONTACTS AND LOCATIONS:
Overall Officials: Abigail Sveden, MS, CGC, Study Chair — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chopra M, McEntagart M, Clayton-Smith J, Platzer K, Shukla A, Girisha KM, Kaur A, Kaur P, Pfundt R, Veenstra-Knol H, Mancini GMS, Cappuccio G, Brunetti-Pierri N, Kortum F, Hempel M, Denecke J, Lehman A; CAUSES Study; Kleefstra T, Stuurman KE, Wilke M, Thompson ML, Bebin EM, Bijlsma EK, Hoffer MJV, Peeters-Scholte C, Slavotinek A, Weiss WA, Yip T, Hodoglugil U, Whittle A, diMonda J, Neira J, Yang S, Kirby A, Pinz H, Lechner R, Sleutels F, Helbig I, McKeown S, Helbig K, Willaert R, Juusola J, Semotok J, Hadonou M, Short J; Genomics England Research Consortium; Yachelevich N, Lala S, Fernandez-Jaen A, Pelayo JP, Klockner C, Kamphausen SB, Abou Jamra R, Arelin M, Innes AM, Niskakoski A, Amin S, Williams M, Evans J, Smithson S, Smedley D, de Burca A, Kini U, Delatycki MB, Gallacher L, Yeung A, Pais L, Field M, Martin E, Charles P, Courtin T, Keren B, Iascone M, Cereda A, Poke G, Abadie V, Chalouhi C, Parthasarathy P, Halliday BJ, Robertson SP, Lyonnet S, Amiel J, Gordon CT. Heterozygous ANKRD17 loss-of-function variants cause a syndrome with intellectual disability, speech delay, and dysmorphism. Am J Hum Genet. 2021 Jun 3;108(6):1138-1150. doi: 10.1016/j.ajhg.2021.04.007. Epub 2021 Apr 27. PMID 33909992